CLINICAL TRIAL: NCT00437983
Title: A Single-Center, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy of Phosphatidylserine-Omega3 in Elderly With Age Associated Memory Impairment
Brief Title: The Efficacy of Phosphatidylserine-Omega3 in Elderly With Age Associated Memory Impairment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Enzymotec (Industry)
Responsible Party: Yael Richter PhD, Enzymotec
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Memory_PS 001
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Results first posted 2009-11-25 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2010-01

CONDITIONS: Age Associated Memory Impairment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- PS-Omega3 (Active Comparator): Phosphatidylserine-Omega3, 300mg/day 15 wk
  Interventions: Dietary Supplement: PS-Omega3
- Placebo (Placebo Comparator): Cellulose tainted with fishy odor, 3 capsules/day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: PS-Omega3 — Phosphatidylserine-Omega3 capsules 3x100mg/day 15 wk. Next, follow up phase, open label,1x100mg/day, 15 wk
  Arms: PS-Omega3
Dietary Supplement: Placebo — Placebo cellulose tainted with fishy odor capsules 3x100mg/day 15 wk
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to assess the ability of an oral administration of Phosphatidylserine-Omega3 to improve attention and memory complaints in comparison to placebo in age associated memory impaired subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give written informed consent
2. Age: 90≥ years ≥50
3. Gender: male and female
4. CDR ≤ 0.5
5. Complaints of memory loss reflected in such everyday problems as difficulty remembering names of individuals following introduction, misplacing objects, difficulty remembering multiple items to be purchased or multiple tasks to be performed, difficulty remembering telephone numbers or zip codes, and difficulty recalling information quickly or following distraction. Onset of memory loss must be described as gradual, without sudden worsening in recent months. Complaints of memory loss to be assessed by the MAC-Q scale.
6. Mini-Mental State Examination (MMSE) ≥27 for subjects with college education (BA) and ≥ 26 for all others
7. Memory test performance that is at least 1 SD below the mean established for young adults on at least one neuropsychological subtest of NexAde.
8. Language: Subjects must be able to read, write and speak Hebrew.
9. Ability to perform tests and interviews

Exclusion Criteria:

1. Evidence of delirium, confusion, or other disturbances of consciousness
2. Any Neurological disorder that could produce cognitive deterioration. Such disorders include AD, Parkinson's disease, stroke, intracranial hemorrhage, local brain lesions including tumors, and normal pressure hydrocephalus
3. History of any infective or inflammatory brain disease including those of viral, fungal, or syphilitic etiologies
4. Evidence of significant cerebral vascular pathology
5. Head injury immediately preceding cognitive deterioration.
6. Current psychiatric diagnosis according to DSM IV criteria of depression, mania, or any other major psychiatric disorder
7. Current diagnosis or history of alcoholism or drug dependence.
8. Evidence of depression as determined by the Geriatric Depression Scale (short version) score of 5 or more.
9. Any medical disorder that could produce cognitive deterioration including renal, respiratory, cardiac, and hepatic disease, diabetes mellitus, endocrine, metabolic or hematological disturbances unless well controlled, and malignancy not in remission for more than two years
10. Use of psychotropic drug or any other drug or supplement that may significantly affect cognitive functioning during the month prior to psychometric testing.
11. Use of any experimental medication within 1 month prior to screening or as concomitant medications.
12. Subject has a history of hypersensitivity or allergy to fish or fish oil or soy.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2007-04; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amos Korczyn, MD, Study Director — Sourasky Medical Center
Locations (1):
- The Tel Aviv Sourasky Medical Center, Neurology department, Tel Aviv, Israel

REFERENCES:
- [Derived] Vakhapova V, Richter Y, Cohen T, Herzog Y, Korczyn AD. Safety of phosphatidylserine containing omega-3 fatty acids in non-demented elderly: a double-blind placebo-controlled trial followed by an open-label extension. BMC Neurol. 2011 Jun 28;11:79. doi: 10.1186/1471-2377-11-79. PMID 21711517

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through advertisements in senior citizens' homes, hospitals, and newspapers.
Groups:
- Placebo: Cellulose tainted with fishy odor
Period: Overall Study
Arm/Group | PS-Omega3 | Placebo
Started | 79 | 78
Completed | 66 | 65
Not Completed | 13 | 13
Not completed — Adverse Event | 6 | 6
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PS-Omega3 | Placebo | Total
Number analyzed (Participants) | 79 | 78 | 157
Age Continuous [Mean (Standard Deviation); unit: years] | 72.58 (8.12) | 72.46 (8.33) | 72.52 (8.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 39 | 78
  Male | 40 | 39 | 79
Region of Enrollment [Number; unit: participants]
  Israel | 79 | 78 | 157

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Rey Auditory Verbal Learning Test
Description: A widely used, brief, easy to understand scale to evaluate verbal learning and memory. The score is presented as the number of words correctly recalled (0 is worse, 15 is best).The total learning task score ranges from 0 to 45 words(0 is worse, 45 is best).
Time Frame: baseline, 15 wk
Population: Analysis of per-protocol (PP) cohort. Out of the 131 participants who completed the study, nine were excluded from the PP analysis (5 from the placebo group and 4 from the PS-omega3 group), one due to short interval between visits and the rest didn't meet the compliance criteria (≥ 65%).
Measure: Mean (Standard Error); unit: number of words correctly recalled
Arm/Group | PS-Omega3 | Placebo
Number analyzed (Participants) | 60 | 62
number of words correctly recalled
  Immediate recall | 1.53 (0.26) | 1.00 (0.20)
  Total Learning | 5.30 (0.89) | 4.02 (0.85)
  Delayed recall | 0.93 (0.29) | 0.79 (0.35)

2. Secondary Outcome: Blood Work
Time Frame: baseline,15 wk
Reporting Status: Not Posted

3. Secondary Outcome: Trail Making Test
Time Frame: Baseline, 15 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Computerized Cognitive Assessment Tool
Time Frame: baseline, 15 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Clinical Global Impression of Change (CGI-C)Scale
Description: The Clinical Global Impression of Change (CGI-C)scale is designed to record the clinician's global impression of change. Global improvement score ranges from 1 = "Very much improved", through 4 = "No change", to 7 = "Very much worse". Participants who experienced an improvement (scores 1, 2 or 3) in at least one of the two visits (following 7 or 15 weeks of treatment) were classified as improved over the treatment period (with the exception of participants reporting improvement following 7 weeks and deterioration at endpoint, who were NOT rated as improved)
Time Frame: 7 weeks, 15 weeks
Population: as for outcome 1
Measure: Number; unit: Participants who experienced improvement
Arm/Group | PS-Omega3 | Placebo
Number analyzed (Participants) | 60 | 62
Participants who experienced improvement | 22 | 17

6. Secondary Outcome: Change From Baseline in Rey Osterrieth Complex Figure Test
Description: A widely used neuropsychological tool for the evaluation of visuospatial constructional ability and visual memory. Both the time to complete the task (copy time)and the accuracy (immediate and delayed recall) were used as measures for the analysis. Accuracy range score is 0-36 points (0 is worse, 36 is best). Copy time is expressed in seconds (less time to copy indicates better performance).
Time Frame: baseline, 15 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | PS-Omega3 | Placebo
Number analyzed (Participants) | 60 | 62
Units on a scale
  Copy Time (sec) | -23.27 (8.92) | 3.73 (12.44)
  Immediate recall | 2.73 (0.68) | 1.35 (0.66)
  Delayed recall | 2.28 (0.68) | 2.37 (0.67)

ADVERSE EVENTS:
Arm/Group | PS-Omega3 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/78
Other Adverse Events (participants affected / at risk) | 0/79 | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No